CLINICAL TRIAL: NCT04093518
Title: A Randomized Trial Administering Estradiol Patch vs. Placebo Patch as add-on to Antipsychotics in Female Patients Above the Age of 38 With Schizophrenia, Schizoaffective or Schizophreniform Disorder
Brief Title: Estradiol as add-on to Antipsychotics
Acronym: EST-S-02
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tangent Data (Other)
Collaborators: Stanley Medical Research Institute (Other); MediStat Ltd. (Unknown); PCI pharma services (formerly BIOTEC SERVICES INTERNATIONAL LIMITED) (Unknown); S.C. IMUNOTEHNOMED S.R.L. (Unknown); Tangent Data Srl (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EST-S-02
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2019-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Estradiol

STUDY DESIGN:
Intervention Model Description: Randomized, add-on to anti-psychotics, double blind, placebo-controlled, parallel group clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator (Active Comparator): Estradiol 200µg
  Interventions: Drug: Estradiol
- Placebo Comparator (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Estradiol — 2 transdermal patches to be changed twice a week for the duration of 16 weeks
  Other Names: trans dermal patches
  Arms: Active Comparator
Drug: Placebo — 2 transdermal patches to be changed twice a week for the duration of 16 weeks
  Other Names: trans dermal patches
  Arms: Placebo Comparator

SUMMARY:
The objective of the study is to evaluate the efficacy of Estradiol patch compared to placebo, as add-on to anti-psychotics in the treatment of women 38 and older with schizophrenia, schizoaffective or schizophreniform disorder.

DETAILED DESCRIPTION:
Several lines of evidence suggest that estrogen affects the course of schizophrenia. The onset of schizophrenia is 2-4 years later in women than in men, and women have a lower incidence of schizophrenia until menopause, after which women have an increased incidence, so that the lifetime prevalence is similar in both genders. Women are more likely to have their first schizophrenic episode during an estradiol trough in the menstrual cycle. These gender differences in the natural course of schizophrenia are well replicated and provide a major lead to understanding and treating the illness, and have led to several randomized controlled trials administering oral estradiol to patients with schizophrenia. Studies on transdermal estradiol have been more encouraging, and four RCTs, have shown that estradiol patches are efficacious in treating schizophrenia The most recent study was performed our group and showed that overall estradiol patches were efficacious with an effect size of 0.41 for total PANSS, with significant improvements in PANSS positive, negative and general-psychopathology scores. Post hoc analyses showed that the improvements in symptoms were found almost exclusively in women who were 38 and older, in whom the effect of estrogen patches vs placebo reached an effect size of 0.58 for PANSS total.

The currently proposed study is based on the post-hoc finding of improvement in participants aged 38 and above, and we will a-priori recruit women with schizophrenia 38 and above, in order to test the efficacy of 200 µg estradiol patches vs placebo in these woman.

ELIGIBILITY:
Inclusion Criteria:

1. Female above 38, up to 45 years of age, inclusive
2. Willing and able to provide informed consent, after the nature of the study has been fully explained
3. Current DSM-V diagnosis of schizophrenia, schizoaffective or schizophreniform disorder as confirmed by modified SCID.
4. Total PANSS score > 70 and (PANSS positive subscale >15 and/or PANSS negative subscale >15)
5. Must be on a stable dose of any antipsychotic drug, for at least 2 weeks prior to the baseline visit, at doses within the PORT criteria, whenever possible. Patients receiving higher doses will have their records reviewed to ensure that their dose is required and, if possible, will be stabilized on a lower dose prior to study entry.
6. Patients who are physically and endocrinologically healthy,
7. Not menopausal as assessed by asking patients if they are menstruating
8. Inpatients or outpatients. Inpatients will be randomized 3 days or more after admission

Exclusion Criteria:

1. Unwilling or unable, in the opinion of the Investigator, to comply with study instructions
2. Pregnant or breast-feeding
3. Women who are menopausal.
4. Patients treated with oral estrogen preparations containing estradiol greater than 30 mcg.
5. Women who have known severe abnormalities in the hypothalamo-pituitary gonadal axis, thyroid disorders, severe medical conditions and disorders that would contraindicate estrogen use (breast cancer, migraine with aura or stroke)
6. History of endometrial cancer or breast cancer, history of breast or uterine cancer, no history of 1st and 2nd grade family with breast or uterine cancer, vaginal bleeding between periods.
7. Likely allergy or sensitivity to estradiol.
8. Schizoaffective disorder in the manic phase.
9. At significant risk of committing suicide, or in the opinion of the Investigator, currently at imminent risk of suicide or harming others.
10. Patients with a current DSM-V substance or alcohol abuse. Patients with a history of and/or current recreational use of cannabinoids or alcohol, and/or patients who smoke cigarettes can be included.
11. Concurrent delirium, mental retardation, drug-induced psychosis, or history of clinically significant brain trauma documented by CT or MRI.
12. Patients receiving phenobarbital, phenytoin, carbamazepine, rifampicin, rifabutin, nevirapine, efavirenz, ritonavir and nelfinavir,or Hypericum perforatum.

Ages: 38 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Gender identity
Enrollment: 100 (Estimated)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-10-15 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in total PANSS scores at the end of the trial | Change from Baseline at 16 weeks
  The Positive and Negative Syndrome Scale (PANSS) is a well validated, standardized method of evaluating and monitoring psychotic symptoms. The PANSS assesses: positive (hallucinations, delusions, thought disorder), negative (blunted affect, abstract thinking and general symptomatology. The positive and negative subscale each consist of 7 items rated from 1(absent) - 7(extreme) with a minimum score = 7, maximum score = 49. The general subscale consists of 16 items with a minimum score = 16, maximum score = 112. A Total PANSS score (positive+ negative + general scores) has a minimum of 30 and maximum of 210. Higher scores represent more severity in symptoms.

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) and general psychopathology scales | through study, 16 weeks
  To evaluate the effects of Estradiol on Positive and Negative Syndrome Scale (PANSS)
Clinical Global Impression Scale-Severity (CGI-S) and Global Impression Scale-Improvement (CGI-I), | through study, 16 weeks
  To evaluate the effects of Estradiol vs Placebo on Clinical Global Impression
Montgomery-Asberg Depression Rating Scale | through study, 16 weeks
  To evaluate the effects of Estradiol on depressive symptoms
Rates of drop outs before the end of the trial | through study completion, an average of 1 year
  To evaluate the rate of drop outs

CONTACTS AND LOCATIONS:
Overall Officials: Mark Weiser, M.D., Principal Investigator — Sheba Medical Center
Locations (1):
- Centrul Comunitar de Sănătate Mintală Botanica, Chisinau, Moldova

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Angermeyer MC, Kuhn L, Goldstein JM. Gender and the course of schizophrenia: differences in treated outcomes. Schizophr Bull. 1990;16(2):293-307. doi: 10.1093/schbul/16.2.293. PMID 2374885
- [Result] Goff DC, Henderson DC, Amico E. Cigarette smoking in schizophrenia: relationship to psychopathology and medication side effects. Am J Psychiatry. 1992 Sep;149(9):1189-94. doi: 10.1176/ajp.149.9.1189. PMID 1503131
- [Result] Harrison G, Croudace T, Mason P, Glazebrook C, Medley I. Predicting the long-term outcome of schizophrenia. Psychol Med. 1996 Jul;26(4):697-705. doi: 10.1017/s0033291700037715. PMID 8817704
- [Result] Heringa SM, Begemann MJ, Goverde AJ, Sommer IE. Sex hormones and oxytocin augmentation strategies in schizophrenia: A quantitative review. Schizophr Res. 2015 Nov;168(3):603-13. doi: 10.1016/j.schres.2015.04.002. Epub 2015 Apr 23. PMID 25914107
- [Result] Jeste DV, Lindamer LA, Evans J, Lacro JP. Relationship of ethnicity and gender to schizophrenia and pharmacology of neuroleptics. Psychopharmacol Bull. 1996;32(2):243-51. PMID 8783894
- [Result] Kulkarni J, Gavrilidis E, Worsley R, Hayes E. Role of estrogen treatment in the management of schizophrenia. CNS Drugs. 2012 Jul 1;26(7):549-57. doi: 10.2165/11630660-000000000-00000. PMID 22626057
- [Result] Magharious W, Goff DC, Amico E. Relationship of gender and menstrual status to symptoms and medication side effects in patients with schizophrenia. Psychiatry Res. 1998 Feb 27;77(3):159-66. doi: 10.1016/s0165-1781(97)00137-6. PMID 9707298
- [Result] Melkersson KI, Hulting AL, Rane AJ. Dose requirement and prolactin elevation of antipsychotics in male and female patients with schizophrenia or related psychoses. Br J Clin Pharmacol. 2001 Apr;51(4):317-24. doi: 10.1046/j.1365-2125.2001.01352.x. PMID 11318766
- [Result] Opjordsmoen S. Long-term clinical outcome of schizophrenia with special reference to gender differences. Acta Psychiatr Scand. 1991 Apr;83(4):307-13. doi: 10.1111/j.1600-0447.1991.tb05545.x. PMID 2028808
- [Result] Pardridge WM, Mietus LJ. Transport of steroid hormones through the rat blood-brain barrier. Primary role of albumin-bound hormone. J Clin Invest. 1979 Jul;64(1):145-54. doi: 10.1172/JCI109433. PMID 447850
- [Result] Pinals DA, Malhotra AK, Missar CD, Pickar D, Breier A. Lack of gender differences in neuroleptic response in patients with schizophrenia. Schizophr Res. 1996 Dec 15;22(3):215-22. doi: 10.1016/s0920-9964(96)00067-9. PMID 9000318
- [Result] Seeman MV. Gender differences in the prescribing of antipsychotic drugs. Am J Psychiatry. 2004 Aug;161(8):1324-33. doi: 10.1176/appi.ajp.161.8.1324. PMID 15285956
- [Result] Szymanski S, Lieberman JA, Alvir JM, Mayerhoff D, Loebel A, Geisler S, Chakos M, Koreen A, Jody D, Kane J, et al. Gender differences in onset of illness, treatment response, course, and biologic indexes in first-episode schizophrenic patients. Am J Psychiatry. 1995 May;152(5):698-703. doi: 10.1176/ajp.152.5.698. PMID 7726309
- [Result] Torgalsboen AK. Full recovery from schizophrenia: the prognostic role of premorbid adjustment, symptoms at first admission, precipitating events and gender. Psychiatry Res. 1999 Nov 8;88(2):143-52. doi: 10.1016/s0165-1781(99)00077-3. PMID 10622350
- [Result] Usall J, Araya S, Ochoa S, Busquets E, Gost A, Marquez M; Assessment Research Group in Schizophrenia (NEDES). Gender differences in a sample of schizophrenic outpatients. Compr Psychiatry. 2001 Jul-Aug;42(4):301-5. doi: 10.1053/comp.2001.24582. PMID 11458304
- [Result] an der Heiden W, Krumm B, Muller S, Weber I, Biehl H, Schafer M. [The Mannheim long-term study of schizophrenia. Initial results of follow-up of the illness over 14 years after initial inpatient treatment]. Nervenarzt. 1995 Nov;66(11):820-7. German. PMID 8532098
- [Result] van der Werf M, Hanssen M, Kohler S, Verkaaik M, Verhey FR; RISE Investigators; van Winkel R, van Os J, Allardyce J. Systematic review and collaborative recalculation of 133,693 incident cases of schizophrenia. Psychol Med. 2014 Jan;44(1):9-16. doi: 10.1017/S0033291712002796. Epub 2012 Dec 17. PMID 23244442